CLINICAL TRIAL: NCT00934765
Title: Effect of Weight Loss on Reproductive Function in Overweight Men.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University College (Other)
Collaborators: Oslo University Hospital (Other); The Hospital of Vestfold (Other); Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Oliwia Witczak, associate professor, Oslo Metropolitan University
Other Study IDs: HiO 08/220b
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Overweight; Obesity
Keywords: overweight, obesity, male, fertility
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, semen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: weight loss — self-directed weight loss, guided weight loss, weight loss by gastric by-pass surgery

SUMMARY:
Obesity has been found to be a risk factor for female infertility. Studies have indicated that obese men often have poor semen quality and require increased time to make partner pregnant. To date, no studies have investigated the effect of weight reduction on male fertility. The purpose of this study is to investigate the effect of weight reduction in overweight and obese men on their reproductive function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* BMI > 27 kg/m2

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese and overweight men that are planing to loss weight by diet and/or lifestyle changes or gastric by-pass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-09; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
weight, height, % body fat, sperm (volume, concentration, motility, morphology, vitality), sperm DNA integrity, steroid hormones, gonadotropins, blood glucose, HbA1c, mCRP, lipids, adiponectins, fatty acid composition in serum and sperm phospholipids | minimum three months

SECONDARY OUTCOMES:
genetic variations in genes involved in metabolism and reproduction | no time frame

CONTACTS AND LOCATIONS:
Overall Officials: Trine B. Haugen, PhD, Study Chair — Oslo University College; Oliwia Witczak, PhD, Principal Investigator — Oslo University College
Locations (1):
- Oslo University College, Oslo, Norway